CLINICAL TRIAL: NCT02324478
Title: Exploration of Autonomic Nervous System by Photoplethysmography
Status: Completed | Type: Observational
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Riccardo Colombo, autonomic nervous system analysis during laparoscopy, ASST Fatebenefratelli Sacco
Other Study IDs: ANSSi_2
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Intervention Affecting Autonomic Nervous System
Keywords: autonomic nervous system; heart rate variability; laparoscopic surgery; general anesthesia; photoplethysmography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: autonomic nervous system analysis — electrocardiographic and pulse-photoplethysmographic waves of patients under general anesthesia for laparoscopic cholecystectomy will be recorded on a laptop pc for offline analysis of autonomic nervous system modulation a three main time point: 1) at baseline, before general anesthesia induction, 2) five min after tracheal tube placement, 3) five min after pneumoperitoneum insufflation.

SUMMARY:
The autonomic nervous system state (ANSS) and the autonomic nervous system state index (ANSSi) - two indices derived from the pulse photo-plethysmography analysis - have been recently advocated as a measure of sympathetic activity in the anesthetized patients, but their validity has not been yet demonstrated. We will conduct a study aiming to assess if ANSS and ANSSi reflect autonomic nervous system modulation on cardiovascular system in healthy humans under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 50 years
* American Society of Anaesthesiologists status I and II

Exclusion Criteria:

* hypertension requiring pharmacological treatment or chronic cardiovascular disease
* arrhythmic cardiac disease (atrial fibrillation, atrial flutter, ectopic beats >5% of normal sinus beats)
* history of alcohol or drug abuse
* obesity (BMI>30)
* diabetes or other endocrine pathology (thyroidal or adrenal)
* peripheral neuropathy or any kind of chronic neurological disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adults scheduled for elective laparoscopic cholecystectomy under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
autonomic nervous system activity during laparoscopic cholecystectomy (measured by pulse-photoplethysmography and heart rate variability analysis) | 120 min
  assessment of autonomic nervous system activity measured by pulse-photoplethysmography and heart rate variability analysis

SECONDARY OUTCOMES:
agreement of photoplethysmography and heart rate variability | 120 min
  assessment of agreement between pulse-photoplethysmography and heart rate variability as a measure of autonomic nervous system activity

CONTACTS AND LOCATIONS:
Locations (1):
- Luigi Sacco Hospital, Milan, Italy

REFERENCES:
- [Background] Hamunen K, Kontinen V, Hakala E, Talke P, Paloheimo M, Kalso E. Effect of pain on autonomic nervous system indices derived from photoplethysmography in healthy volunteers. Br J Anaesth. 2012 May;108(5):838-44. doi: 10.1093/bja/aes001. Epub 2012 Feb 26. PMID 22369767
- [Background] Colombo R, Raimondi F, Corona A, Rivetti I, Pagani F, Porta VD, Guzzetti S. Comparison of the Surgical Pleth Index with autonomic nervous system modulation on cardiac activity during general anaesthesia: A randomised cross-over study. Eur J Anaesthesiol. 2014 Feb;31(2):76-84. doi: 10.1097/01.EJA.0000436116.06728.b3. PMID 24284309
- [Background] Sly WS, Sato S, Zhu XL. Evaluation of carbonic anhydrase isozymes in disorders involving osteopetrosis and/or renal tubular acidosis. Clin Biochem. 1991 Aug;24(4):311-8. doi: 10.1016/0009-9120(91)80005-n. PMID 1959222
- [Background] Monk TG, Ding Y, White PF. Total intravenous anesthesia: effects of opioid versus hypnotic supplementation on autonomic responses and recovery. Anesth Analg. 1992 Nov;75(5):798-804. doi: 10.1213/00000539-199211000-00026. PMID 1358002
- [Background] Myles PS, Cui J. Using the Bland-Altman method to measure agreement with repeated measures. Br J Anaesth. 2007 Sep;99(3):309-11. doi: 10.1093/bja/aem214. No abstract available. PMID 17702826
- [Background] O'Leary E, Hubbard K, Tormey W, Cunningham AJ. Laparoscopic cholecystectomy: haemodynamic and neuroendocrine responses after pneumoperitoneum and changes in position. Br J Anaesth. 1996 May;76(5):640-4. doi: 10.1093/bja/76.5.640. PMID 8688262
- [Background] Paloheimo MP, Sahanne S, Uutela KH. Autonomic nervous system state: the effect of general anaesthesia and bilateral tonsillectomy after unilateral infiltration of lidocaine. Br J Anaesth. 2010 May;104(5):587-95. doi: 10.1093/bja/aeq065. Epub 2010 Mar 30. PMID 20354006
- [Background] Porta A, Baselli G, Caiani E, Malliani A, Lombardi F, Cerutti S. Quantifying electrocardiogram RT-RR variability interactions. Med Biol Eng Comput. 1998 Jan;36(1):27-34. doi: 10.1007/BF02522854. PMID 9614745